CLINICAL TRIAL: NCT05240547
Title: Chiropractic Spinal Manipulation for Cervicogenic and Tension-type Headache: a Pilot and Feasibility Study
Brief Title: Chiropractic Spinal Manipulation for Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Real Centro Universitario Maria Cristina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMTHA
Record Dates: First submitted 2022-02-01; First posted 2022-02-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cervicogenic Headache; Tension-Type Headache
MeSH Terms: conditions — Post-Traumatic Headache; Tension-Type Headache | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal manipulation (Experimental): Spinal manipulative therapy will be delivered to the cervical spine (segments including occiput-atlas to C7-D1) according to the chiropractors' evaluation during each visit. During each session, one or two segments will be manipulated using a high-velocity low-amplitude thrust manipulation (a joint cavitation will be expected, if not, the thrust can repeated once) applied to the segments with the highest motion restriction, as determined by the chiropractor by static and motion palpation of the cervical spine.
  Interventions: Other: Spinal Manipulation
- Placebo (Placebo Comparator): Sham manipulation will be delivered to the cervical spine (segments including occiput-atlas to C7-D1) according to the chiropractors' evaluation during each visit. During each session, one or two segments will receive a sham manipulation applied to the segments with the highest motion restriction, as determined by the chiropractor by static and motion palpation of the cervical spine. The sham manipulation will consist in a identical contact to the real manipulation, except the thrust will be delivered towards the table, away from the target segment and with the intention to lower the cervical drop piece of the table, which will substitute the joint cavitation noise.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Spinal Manipulation — Spinal manipulative therapy delivered to the cervical spine by a chiropractor
  Arms: Spinal manipulation
Other: Placebo — Sham manipulative treatment delivered to the cervical spine by a chiropractor
  Arms: Placebo

SUMMARY:
This is a pilot and feasibility randomized controlled trial to assess the efficacy of chiropractic spinal manipulative therapy in patients with tension-type and cervicogenic headache.

DETAILED DESCRIPTION:
This study is a pilot and feasibility randomized controlled trial that aims to assess the efficacy of 8 treatment sessions of chiropractic spinal manipulative therapy compared to the same number of sham manipulative therapy or placebo interventions for chronic cervicogenic and tension-type headache. The hypothesis proposed is that chiropractic care will reduce the intensity and frequency of both cervicogenic and tension-type headache episodes, when compared to placebo. A sample of 20 participants suffering from cervicogenic or tension-type headache for at least 3 months, aged 18 to 67 will be randomized to receive either 8 sessions of spinal manipulative treatment (2 times per week for a total of 4 weeks) or 8 sessions of a validated sham spinal manipulation. Outcomes will be assessed at baseline, after 4 treatments and at the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 episodes per month of cervicogenic or tension-type headache for at least 3 months. Diagnoses will be determined by case history and physical examination according to the International Headache Society criteria (3rd Edition)

Exclusion Criteria:

* Not fulfilling the inclusion criteria
* Having received chiropractic treatment in the previous 12 months
* Diagnosis or frequent symptoms of migraine headaches (symptoms present at least once a month) without an overlapping presentation of cervicogenic or tension-type headache.
* Patients with pathologies affecting the nervous system (MS, tumors, past history of stroke...)
* Contraindications to manual therapy, particularly spinal manipulative therapy (cancer, uncontrolled high blood-pressure, severe cardiovascular conditions)
* Past history of cervical spine surgery
* Pregnancy
* Having being diagnosed with a psychiatric conditions, with the exception of depression and anxiety

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Pain intensity will be measured by showing patients a numerical rating scale from 0 (no pain at all) to 10 (maximum possible pain)
Pain frequency | 4 weeks
  Chronic pain patients will describe whether their pain is episodic (pain-free periods of at least 4 week duration) or fluctuating (no pain-free periods of at least 4 week duration)

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | 4 weeks
  The Pain Catastrophizing Scale (PCS) provides the level of catastrophizing beliefs and emotions that a person has with regards to his/her own pain experience, in this case, low back pain. It includes 13 items rated on a Likert scale from 0-4. The total range of possible scores is from 0-52, where 0 is the lowest possible level of catastrophizing and 52 the highest.
Pressure pain thresholds | 4 weeks
  Pressure pain thresholds (PPTs) are part of quantitative sensory testing. The aim is to identify the threshold and the sensitivity to suprathreshold pressure stimulation in different areas of the patients' bodies. An algometer will be used (Wagner Force Dial FDK20, Greenwich, CT, USA) to measure PPTs in the suboccipital muscles for each patient. The measure will be taken before and after treatment to determine the immediate effects of spinal manipulative therapy on pain sensitivity. this will be used to correlate with the changes in clinical pain.

OTHER OUTCOMES:
Sex | 4 months
  Biological sex (Male or Female) for feasibility purposes
Age | 4 months
  Age (measured in years) for feasibility purposes
Costs for care | 4 months
  The costs related to the time dedicated by researchers to the study will be calculated in Euros.
Costs in stipends | 4 months
  Costs per participant for care received will be calculated in Euros.
Total number of potential participants recruited initially | 4 months
  The total number of participants recruited at the beginning of the study will be recorded as an outcome in order to calculate Drop-out ratios (dividing the number of participants completing the study by the total number of initially recruited).
Total number of potential participants who made contact showing an interest in the study | 4 months
  The total number of potential participants interested in the study will be recorded as an outcome in order to calculate Recruitment ratio (dividing the number of participants initiating the study by the total number of interested).
Total number of participants completing the study | 4 months
  The number of participants recruited and completing the study will be recorded as an outcome to be later divided by the number of months of the study, in order to calculate the recruitment rate.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gevers Montoro, DC, MSc, Principal Investigator — RCU María Cristina
Locations (1):
- Real Centro Universitario María Cristina, El Escorial, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No